CLINICAL TRIAL: NCT01153724
Title: Relative Bioavailability of 10 mcg Olodaterol (Solution for Inhalation Administered With the Respimat) at Steady State Alone or in Combination With Multiple Doses of 400 mg q.d. Fluconazole (Hard Capsule) in Healthy Male and Female Volunteers (an Open Label, Fixed Sequence, Phase I Study)
Brief Title: Relative Bioavailability of Olodaterol and Fluconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222.48; 2010-018528-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-05

CONDITIONS: Healthy; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Fluconazole

ARMS (2):
- Olodaterol (Experimental)
  Interventions: Drug: BI 1744
- Olodaterol + Fluconazole (Experimental)
  Interventions: Drug: BI 1744; Drug: Fluconazole

INTERVENTIONS:
Drug: BI 1744 — 10 mcg solution for oral inhalation
Drug: Fluconazole — 400 mg capsule
  Arms: Olodaterol + Fluconazole

SUMMARY:
This clinical trial is intended to investigate a possible effect of the CYP 2C9 inhibitor fluconazole on the bioavailability of olodaterol

ELIGIBILITY:
Inclusion criteria:

Healthy male and female volunteers

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1222.48.1 Boehringer Ingelheim Investigational Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Total number of patients treated in the study. This was an open-label, fixed sequence, phase I trial in healthy volunteers. 35 subjects received in period 1 Olodaterol 10 microgram delivered by Respimat inhaler once daily for 8 days and in period 2 Olodaterol 10 microgram delivered by Respimat inhaler once daily plus 1 capsule Fluconazole 400 milligram once daily, both for 14 days (with a loading dose of 800 milligram on the first day).
Period: Treatment Period 1
Arm/Group | Overall Study
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment Period 2
Arm/Group | Overall Study
Started | 34
Completed | 32
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Other reason not defined above | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve From 0 to 6 Hours at Steady State (AUC0-6,ss)
Description: AUC0-6,ss represents the area under the concentration curve of olodaterol in plasma from 0 to time t=6 hours at steady state, where t is defined as the latest time-point where at least 2/3 of the subjects in both treatment periods reveal quantifiable plasma concentrations of olodaterol. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: Pharmacokinetic (PK) analysis set includes all evaluable subjects in the treated set providing at least 1 observation for at least 1 PK endpoint without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Groups:
- Olodaterol: Oral inhalation of Olodaterol 10 microgram solution with Respimat A5 device once daily for 8 days.
- Olodaterol Plus Fluconazole: Oral inhalation of Olodaterol 10 microgram solution with Respimat A5 device once daily for 14 days plus Fluconazole 400mg capsule administered orally once daily for 14 days.
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 24 | 28
Picogram*hours/milliliter | 19.659 (13.6) | 22.271 (13.6)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Fluconazole; Ratio Olodaterol plus Fluconazole and Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0101, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 113.29, 90% CI 2-sided [105.893 to 121.197], Standard Deviation 13.6 — The standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Maximum Concentration at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum concentration of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma at steady state. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 33 | 32
Picogram/milliliter
  Olodaterol (N=30;32) | 5.336 (15.5) | 5.805 (15.5)
  Olodaterol glucuronide (N=33;32) | 4.211 (19.4) | 3.621 (19.4)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Fluconazole; Ratio Olodaterol plus Fluconazole and Olodaterol for the category Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0009, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 108.78, 90% CI 2-sided [101.590 to 116.487], Standard Deviation 15.5 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Olodaterol vs Olodaterol Plus Fluconazole; Ratio Olodaterol plus Fluconazole and Olodaterol for the category Olodaterol glucuronide; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0711, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean = 85.98, 90% CI 2-sided [79.277 to 93.253], Standard Deviation 19.4 — The standard deviation is actually the geometric coefficient of variation

3. Secondary Outcome: Time From Dosing to the Maximum Concentration at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to maximum concentration of olodaterol and olodaterol glucuronide in plasma at steady state.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 33 | 32
Hours
  Olodaterol (N=30;32) | 0.250 [0.117 to 1.00] | 0.250 [0.0830 to 1.00]
  Olodaterol glucuronide (N=33;32) | 2.00 [0.0330 to 22.9] | 2.03 [0.0330 to 23.0]

4. Secondary Outcome: Fraction of Urine Excretion From 0 to 24 Hours at Steady State (fe0-24,ss)
Description: fe0-24,ss represents the fraction of olodaterol eliminated in urine from time point 0 to 24 hours after administration at steady state.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of olodaterol
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 32 | 32
percentage of olodaterol | 5.63 (39.8) | 6.45 (33.1)

5. Secondary Outcome: Amount of the Analyte Excreted in Urine From 0 to 24 Hours at Steady State (Ae0-24,ss)
Description: Ae0-24,ss represents the amount of olodaterol and olodaterol glucuronide excreted in urine from 0 to time t=24 at steady state. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 32 | 32
ng
  Olodaterol | 563.459 (33.5) | 647.004 (33.5)
  Olodaterol glucuronide | 465.946 (26.5) | 347.030 (26.5)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Fluconazole; Ratio Olodaterol plus Fluconazole and Olodaterol for the category Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.1539, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 114.83, 90% CI 2-sided [99.940 to 131.932], Standard Deviation 33.5 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Olodaterol vs Olodaterol Plus Fluconazole; Ratio Olodaterol plus Fluconazole and Olodaterol for the category Olodaterol glucuronide; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.8574, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 74.48, 90% CI 2-sided [66.619 to 83.266], Standard Deviation 1.068 — The standard deviation is actually the geometric coefficient of variation

6. Secondary Outcome: Area Under Curve From 0 to 12 Hours at Steady State (AUC0-12,ss)
Description: AUC0-12,ss represents the area under the concentration curve of olodaterol glucuronide in plasma from 0 to time t=12 at steady state, where t is defined as the latest timepoint where at least 2/3 of the subjects in both treatment periods reveal quantifiable plasma concentrations of the analyte. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 27 | 29
Picogram*hours/milliliter | 33.389 (14.6) | 24.735 (14.6)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Fluconazole; Ratio Olodaterol plus Fluconazole and Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.9646, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 74.08, 90% CI 2-sided [69.105 to 79.418], Standard Deviation 14.6 — The standard deviation is actually the geometric coefficient of variation

7. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: First administration of trial medication until 6 days after last administration of trial medication
Population: Treated set (TS) - Treated set includes all patients who had taken at least 1 dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 35 | 34
participants | 0 | 0

8. Secondary Outcome: Assessment of Tolerability by the Investigator
Description: The investigator assessed tolerability based on adverse events and the laboratory evaluation at the end-of-trial examination. The investigator classified the overall tolerability according to the categories 'good', 'satisfactory', 'not satisfactory', and 'bad'.
Time Frame: End of period 1 and end of period 2
Population: TS
Measure: Number; unit: participants
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Number analyzed (Participants) | 35 | 34
participants
  Good | 35 | 30
  Satisfactory | 0 | 3
  Not satisfactory | 0 | 0
  Bad | 0 | 1
  Not assessable | 0 | 0

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 6 days after last administration of trial medication
Description: Adverse events presented for treated set which includes all patients who had taken at least 1 dose of trial medication.
Arm/Group | Olodaterol | Olodaterol Plus Fluconazole
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 2/35 | 18/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (N=35) | Olodaterol Plus Fluconazole (N=34)
Constipation (Gastrointestinal disorders) | 1 | 2
Paraesthesia oral (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 0 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9
Headache (Nervous system disorders) | 1 | 5
Sleep disorder (Psychiatric disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes